CLINICAL TRIAL: NCT03963609
Title: Multi-slice CT Coronary Angiography Assessment of Remodeling Index in Patients With Low to Intermediate Risk Stable Angina
Brief Title: Multi-slice CT Coronary Angiography in Patients With Stable Angina
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, shaimaa Mostafa, assistant professor, Benha University
Other Study IDs: 1258ase
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Chronic Stable Angina
Keywords: chronic stable angina; multislice CT; remodeling index
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: multisclice CT — assessment of the remodeling index by multisclice CT in patients with chronic stable angina

SUMMARY:
early identification of vulnerable plaques by remodeling index prior to rupture and development of acute event is of considerable importance especially by a reliable non-invasive method as CT coronary angiography.

DETAILED DESCRIPTION:
single-center, cross section, observational study included 150 patients with stable angina with normal resting ECG, negative markers, normal systolic function by 2D echocardiography (EF>50%) and without regional wall motion abnormality at rest who were referred to MSCT evaluation of the coronary artery tree.

ELIGIBILITY:
Inclusion Criteria:

* first attack, low to intermediate risk stable angina
* normal resting ECG,
* negative markers
* normal systolic function by 2D echocardiography (EF>50%)
* without regional wall motion abnormality at rest who were referred to MSCT evaluation of the coronary artery tree.

Exclusion Criteria:

* previous acute coronary syndrome or revascularization, those with renal impairment or dye hypersensitivity, patients with morbid obesity (BMI>40kg/m²), rhythm other than sinus rhythm inability to hold breath for 10sec to acquire the image lesions with heavy calcium score.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: evaluation of coronary artery remodeling index in patients with low to intermediate risk stable angina by MSCT coronary angiography.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
remodeling of the coronary artery | 2 years
  to study the changes in wall of the arteries in patients with chronic stable angina early changes don't appear in coronary angiography as it occurs in the form of positive remodeling which can be detected by multisclice coronary angiography Remodeling index is defined as the ratio of the maximum vessel area (or diameter) to a normal reference vessel area (or diameter), and plaques are classified as having significant positive remodeling when the remodeling index is >1.1

REFERENCES:
- [Derived] Mostafa SA, Aboelazem T, Sanad O, Abdelghafar H, Azam A. Multi-slice CT coronary angiography assessment of remodeling index in patients with low- to intermediate-risk stable angina. Egypt Heart J. 2019 Sep 11;71(1):7. doi: 10.1186/s43044-019-0011-5. PMID 31659543